CLINICAL TRIAL: NCT00388739
Title: Initiation of Chronic Asthma Care Regimens in the Pediatric Emergency Department
Acronym: IRUSBUPR0045
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Different study was designed
Sponsor: Baylor College of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Andrea Cruz, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-19489
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Pediatric Asthma; Pulmicort; TEDAS ED; Acute exacerbation of asthma; Chronic asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Albuterol; Prednisolone

STUDY DESIGN:
Intervention Model Description: This was a health outcomes intervention trial that utilized a randomized clinical trial (non-placebo controlled) with two separate arms. All patients received steroids and bronchodilators, but then were randomized to either no intervention or to Pulmicort respules
Masking Description: patients will be randomized to a control and intervention group. Randomization will occur utilizing assignment by a randomized number table. The randomization scheme will then be packaged into sealed envelopes concealed to the educational interventionist at the time of enrollment. Once the patient is enrolled, the interventionist will open the sealed envelope revealing assignment to intervention or control.

ARMS (2):
- Usual care (Active Comparator): Systemic steroids (4 days of prednisone, 1mg/kg/dose to a maximum of 40 mg/dose to be given twice a day). Subjects will also receive standardized discharge medication instructions for using albuterol nebulizer treatments: they will receive a prescription for 2.5mg of albuterol in 3cc Normal Saline for aerosol use via compressor every 3 times a day as a chronic care regimen if they are either in the treatment arm and 1-5 years of age or if they are in the control group and already own a nebulization compressor. Children in the control group that do not own a nebulization compressor will be given a prescription for an albuterol MDI with mask and spacer with instructions to deliver 2 puffs (90mcg per actuation) 3 times a day as a standard chronic care regimen. Instructions to follow-up with their primary care physician in 3-5 days (as is standard care practice) will be given at discharge for patients in the control or treatment arm.
  Interventions: Drug: Usual care: albuterol + systemic steroids
- Usual care + 6 months of inhaled steroids (Experimental): In addition to the usual care described above, patients randomized to the intervention/experimental arm will also be given a one month supply as well as a prescription (for a 6 month supply) for Budesonide respules (children with mild persistent disease will receive 0.25 mg bid whereas children with moderate or severe persistent disease will receive 0.5 mg bid).
  Interventions: Drug: Intervention: Budesonide; Drug: Usual care: albuterol + systemic steroids

INTERVENTIONS:
Drug: Intervention: Budesonide — Patients 1-5 years of age who are randomly assigned to the treatment arm will be given a one month supply as well as a prescription (for a 6 month supply) for Pulmicort respules (children with mild persistent disease will receive 0.25 mg bid whereas children with moderate or severe persistent disease will receive 0.5 mg bid).
  Other Names: Pulmicort
  Arms: Usual care + 6 months of inhaled steroids
Drug: Usual care: albuterol + systemic steroids — All children (control and treatment arm) will be given a burst dose of steroids (4 days of prednisone, 1mg/kg/dose to a maximum of 40 mg/dose to be given twice a day) at discharge from the ED. All children 1-5 years of age will also receive standardized discharge medication instructions for using albuterol nebulizer treatments: they will receive a prescription for 2.5mg of albuterol in 3cc Normal Saline for aerosol use via compressor every 3 times a day as a chronic care regimen if they are either in the treatment arm and 1-5 years of age or if they are in the control group and already own a nebulization compressor.
  Other Names: Albuterol + prednisolone

SUMMARY:
Hypothesis: Initiating chronic management treatment plans in conjunction with an asthma educational intervention in the pediatric Emergency Department (ED) with anti-inflammatory medication will result in an improvement of ED revisits (and unscheduled return visits). Chronic management intitiation in conjunction with an asthma educational intervention in the pediatric ED with anti-inflammatory medication will also result in improved Quality of Life measure.

Specific aims: 1. To demonstrate that the initiation controller medication therapy in conjunction with asthma education will result in:

1. Decreased return ED visits (or unscheduled primary care physician visits) as compared to a control group over a 12 month period
2. Improved Quality of Life as measured by Bukstein's ITG Quality of Life measure.

   2. To describe the relationship of the initiation of controller medication therapy in conjunction with asthma education with well child visits, missed school/daycare days and behavioral capabilities.

   Objective: To determine the impact of beginning chronic asthma medication regimens after an educational intervention in the ED in pediatric patients 1-18 years of age with mild to moderate persistent asthma.

   Long-term goal/purpose: To demonstrate the success of a model of care that utilizes the emergency department physician to initiate National Asthma Education and Prevention Program (NAEPP) guided chronic asthma therapy in children 1-18 years of age. This model will attempt to bridge the gap in initiation of chronic asthma therapy currently left by a failure of both emergency department and primary care physicians.

DETAILED DESCRIPTION:
This study is a health outcomes intervention trial that utilizes a randomized clinical trial (non-placebo controlled) with two separate arms. The study will be conducted in the ED of Texas Children's Hospital, a tertiary care facility that evaluates over 80,000 children per year. IRB approval has been obtained, and guardians of patients 1-18 years of age will be consented for enrollment. All children will receive standardized burst steroids and broncholdilators (albuterol), however, patients will be randomized to a control and intervention group. Randomization will occur utilizing assignment by a randomized number table. The randomization scheme will then be packaged into sealed envelopes concealed to the educational interventionist at the time of enrollment. Once the patient is enrolled, the interventionist will open the sealed envelope revealing assignment to intervention or control. The study will utilize a post hoc analysis of age subgroups (1 through 5 years of age and 6 through 18 years of age).

Inclusion Criteria:

The enrollees involved must be a child who is 1-18 years of age, with a diagnosis of persistent asthma or reactive airway disease and no other cardiovascular or pulmonary disease not currently on the NAEPP recommended chronic care regimen for controller medication therapy.

Exclusion Criteria:

Patients without a physician's confirmed diagnosis of asthma. Children with concurrent cardiovascular or pulmonary disease. Patients will also be excluded if they do not speak English or Spanish as their primary language.

Eligibility. Any child with a diagnosis of asthma meeting an inclusion criteria of an acute exacerbation of asthma in the emergency department of Texas Children's Hospital will be considered for this study. The patient's family must use English or Spanish as a first language. This study will draw upon pediatric emergency department physicians currently trained through the Texas Emergency Department Asthma Surveillance project for classification of chronic severity. Any child who has been identified as having mild or moderate or severe persistent chronic asthma will be eligible for the study as long as he/she is not on the NAEPP recommended chronic care regimen. Procedure. Once informed consent is obtained, demographic information will be collected as well as information regarding the severity of the acute disease. As per standard ED asthma educational intervention protocol through the TEDAS intervention project, all patients will undergo asthma education utilizing the TEDAS ED asthma platform. This is a brief 20-30 minute personalized laptop-driven intervention delivered by one of the trained TEDAS interventionists. Patients that are enrolled will be randomly entered into either a treatment or control arm. Control vs intervention arms. All children (control and treatment arm) will be given a burst dose of steroids (4 days of prednisone, 1mg/kg/dose to a maximum of 40 mg/dose to be given twice a day) at discharge from the ED. All children 1-5 years of age will also receive standardized discharge medication instructions for using albuterol nebulizer treatments: they will receive a prescription for 2.5mg of albuterol in 3cc Normal Saline for aerosol use via compressor 3 times a day as a chronic care regimen if they are either in the treatment arm and 1-5 years of age or if they are in the control group and already own a nebulization compressor. Children in the control group that do not own a nebulization compressor will be given a prescription for an albuterol MDI with mask and spacer with instructions to deliver 2 puffs (90mcg per actuation) 3 times a day as a standard chronic care regimen. Instructions to follow-up with their primary care physician in 3-5 days (as is standard care practice) will be given at discharge for patients in the control or treatment arm. Treatment arm for patients 1-5 years of age. Patients 1-5 years of age who are randomly assigned to the treatment arm will be given a one month supply as well as a prescription (for a 6 month supply) for Pulmicort respules (children with mild persistent disease will receive 0.25 mg bid whereas children with moderate or severe persistent disease will receive 0.5 mg bid). Those children 1-5 years of age who do not have a nebulization compressor delivery system at home will be provided one at no cost to the patient as part of the study if randomized to the intervention group. Upon the one month follow-up call after the index ED visit, children who have improved symptoms may have reduced treatment regimens as follows: children with mild persistent disease will decrease therapy to 0.25 mg qd, children with moderate persistent disease will decrease therapy to 0.5mg qd, and children with severe persistent disease will continue on 0.5mg bid dosing of Pulmicort respules. Children with worsening symptoms at one month will be referred back to their primary care physician or emergency department at Texas Children's Hospital for further evaluation. Control vs intervention arms. Children who are 6-18 years of age and randomized to the control group will be given a standardized steroid burst at discharge from the ED as outlined above. Additionally, they will receive standardized discharge medication instructions for using albuterol nebulizer treatments: they will receive a prescription for 2.5mg of albuterol in 3cc Normal Saline for aerosol use via compressor every 3 times a day as a chronic care regimen if they already own a nebulization compressor. Children who are 6-18 years of age and randomized to either the control group or treatment group and do not own a nebulization compressor will be given a prescription for an albuterol MDI with spacer with instructions to deliver 2 puffs (90mcg per actuation) 3 times a day as a standard chronic care regimen. Treatment arm for patients 6-18 years of age. Children who are randomized to the intervention group will receive a Pulmicort TBH (200mcg/puff) with instructions to deliver 1 puff per twice a day for mild persistent disease or 2 puffs twice a day if they are of moderate or severe persistent disease. Instructions to follow-up with their primary care physician in 3-5 days (as is standard care practice) will be given at discharge for patients in the control or treatment arm. Upon the one month follow-up call after the index ED visit, children who have improved symptoms may have reduced treatment regimens as follows: children with mild persistent disease will decrease therapy to Pulmicort TBH (200mcg/puff) 1 puff once per day for mild persistent disease or 2 puffs once per day if they are of moderate persistent disease, but will remain on 2 puffs twice a day if they are of severe persistent disease. Children with worsening symptoms at one month will be referred back to their primary care physician or emergency department at Texas Children's Hospital for further evaluation.

Follow-up. All children (intervention and control groups) will receive follow-up calls at 14 days, and 3, 6, 9 and 12 months. Queries for primary and secondary outcomes will be made. Patients' families will be mailed a gift certificate for a local fast-food restaurant or toy store as a token of gratitude for their time after each follow-up call (5$ per contact for a maximum of $30 of gift certificates). The regimen for phone-follow is outlined in the PI's Educational Intervention Study (Sockrider, et al. Delivering Tailored Asthma Family Education in a Pediatric Emergency Room Setting: A Pilot Study. Pediatrics, in press). The one month re-evaluation is only to ascertain that the drug is being used as per recommended usage (ie as per FDA approved indications). Should the drug be changed by the primary care physician, the patient will be left on the drug prescribed by the primary care physician. It is important to remember, as noted in my previous cover letter, that this is not a trial to test the efficacy of a drug, but an intervention in health outcomes research to evaluate the effect of starting controller medications on health care utilization while assessing asthma outcomes. There will be no need to contact the PCP after one-month as the initital contact with the PCP will include an explanation for decreasing the dose of steroids after the acute excaerbation to the dosing recommended by the NAEPP guidelines after the first month unless the patient is experiencing an acute exacerbation. If the PCP changes the therapy, this will be an important outcome to track as this is both relevant and assures generalibility of the findings. Unlike a drug efficacy trial, this trial is intended to measure the health outcomes of the ED intervention of STARTING chronic care. The additional measures for the one month follow-up only assure the drug is being delivered as per initital ED discussion (to include the stepdown) or as per the PCP recommendations. If the PCP instructs the parent not to change the dose or to alter the dose, then this will be taken as priority and the PCP change in plan will be noted and its impact analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The enrollees involved must be a child who is 1-18 years of age, with a diagnosis of persistent asthma or reactive airway disease and no other cardiovascular or pulmonary disease not currently on the NAEPP recommended chronic care regimen for controller medication therapy.

Exclusion Criteria:

* Patients without a physician's confirmed diagnosis of asthma. Children with concurrent cardiovascular or pulmonary disease. Patients will also be excluded if they do not speak English or Spanish as their primary language.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11-01 (Estimated); Primary Completion 2006-11-01 (Estimated); Study Completion 2006-11-01 (Estimated)

PRIMARY OUTCOMES:
ED and primary care provider utilization | 12 months
  Decreased return ED visits (or unscheduled primary care physician visits) as compared to a control group over a 12 month period will be measured by comparisons of total number of ED visits (and unscheduled PCP visits) in each group

SECONDARY OUTCOMES:
Improved Quality of Life as measured by Bukstein's ITG will utilize the scoring system developed by Bukstein to evaluate individual parameters as well as aggregate scores in the control and intervention group at each of the 3 month intervals. Significan | Measured at 3, 9, and 12 months
  Bukstein's ITG is a validated score to evaluate individual parameters as well as aggregate scores in the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea T Cruz, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States